CLINICAL TRIAL: NCT03894319
Title: Use of Lumbar Motion Monitor (LMM) as a Prognostic Tool to Predict Response to Medial Branch Radiofrequency Ablation After Medial Branch Diagnostic Blocks
Brief Title: Use of Lumbar Motion Monitor to Predict Response to Radiofrequency Ablation After Medial Branch Diagnostic Blocks
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient staff for measurement assessments
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, JayeshVallabh, Assistant Professor- Physical Medicine & Rehabilitation, Ohio State University
Other Study IDs: 2018H0197
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is being performed to determine if adding an objective measurement of back function can assess the success of a commonly performed back injection procedure-lumbar medial branch blocks. Researchers also hope to compare whether those who have objective improvements after lumbar medial branch blocks will also have more successful lumbar medial branch radiofrequency ablation.

DETAILED DESCRIPTION:
The current standard of care to determine the success of lumbar medical branch block(s) (MBB) is highly subjective, even if clinicians were to use validated questionairres. Currently, there are no studies that use a validated objective functional outcome measure to practically and efficiently assess lumbar MBB success prior to radiofrequency ablation (RFA). The addition of a validated objective measure of functional impairment to the current standard of care may help us improve in identifying the patients that will benefit from lumbar RFA. It has the potential to minimize procedures of limited benefit with a significant impact on containing healthcare spending. Additionally, it may further knowledge on how to appropriately select patients without relying on the stringent double block diagnostic technique put forth by the CMS that may exclude patients who could greatly benefit from a lumbar RFA.

As the objective measure the study will use a lumber motion monitor (LMM). The LMM weighs less than 5 pounds and fits on with a shoulder harness and belt. The LMM measures motion in all three directions (forward back, side to side, and twisting) just like the spine. The LMM testing may take up to 30 minutes depending on how many tasks can be performed by the participant and how many practice trials are required. The LMM testing includes bending forward and back to upright as fast as possible; comfortably while maintaining a twist position.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 20 years of age to 70 years of age
* Capable and willing to consent
* Participants literate in English language
* Patients with predominately bilateral axial pain and clinical suspicion of lumbar facet pain.
* Patients who have completed conservative care: physical therapy (PT)

Exclusion Criteria:

* History of drug abuse/ dependency
* History of prior lumbar medial branch block or medial branch radiofrequency ablation
* Changes to analgesic regimen in the last 30 days
* Allergy to lidocaine or bupivacaine local anesthetic
* Illiteracy (English)
* Presence of a clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Predominately radicular pain.
* Patient reported limb pain greater than axial low back pain
* Previous lumbar spine surgery
* Any condition that the principle investigator may disqualify the patient
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients at the Ohio State Comprehensive Spine Center scheduled to undergo lumbar medial branch blockade and possible subsequent radiofrequency ablation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Change in functional performance probability P(n). | collected at time points Day 1; Weeks 2,4, and 6; and Months 3,6, and 9
  The Lumbar Motion Monitor (LMM) is an objective, validated, reproducible and accurate tool to rapidly assess the degree of impairment with a sensitivity and specificity of 92% and 97%, respectively. This device provides a functional measure of trunk range of motion, flexion velocity, extension velocity, flexion acceleration, extension acceleration and compares recordings to a normative database. The LMM is able to provide an overall impairment score known as a "functional performance probability(P(n)).

SECONDARY OUTCOMES:
Change in Numeric Rating Scale for Pain | collected at time points Day 1; Weeks 2,4, and 6; and Months 3,6, and 9
  Validated as a measure of pain. Widely used and mandated through the Department of Veterans Affairs as a pain assessment tool.Use of the NRS for MBB and RFA success is the current post procedure assessment standard of care and widely used nationally and within the Ohio State Spine Center clinics.
PROMIS 29 | collected at time points Day 1; Weeks 2,4, and 6; and Months 3,6, and 9
  The PROMIS® 29 Profile v. 2.0 contains 29 items from 8 domains-Physical Function, Depression, Anxiety, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity. These PROMIS® Physical Function measures have been validated for the assessment of back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jayesh Vallabh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States